CLINICAL TRIAL: NCT02540252
Title: Nutritional Status, Eating Pattern and Inflammation Among Patients With Amputation of the Lower Limb - a Longitudinal Cohort Study
Brief Title: Nutrition and Inflammation Among Patients With Lower Limb Amputation
Acronym: Amp-Nu
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Ove Andersen, Research Director, Hvidovre University Hospital
Other Study IDs: PSJ-2015
Record Dates: First submitted 2015-09-01; First posted 2015-09-03 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Malnutrition; Inflammation
Keywords: Lower Limb Amputation; Nutrition; Eating; Inflammation; Nursing
MeSH Terms: conditions — Malnutrition; Inflammation | interventions — Metabolic Networks and Pathways

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum and plasma samples; peripheral blood mononuclear cells (PBMCs); and muscle biopsies
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Nutritional status among patients with lower limb amputation — Patients nutritional status, inflammatory and metabolic pathway are observed during their hospitalization.
  Other Names: Inflammation and metabolic pathway

SUMMARY:
Patients with non-traumatic lower limb amputation are characterized by; high age; majority being men; multimorbidity; and high mortality. The patients comorbidities are related to diabetes and cardiovascular disorders such as arteriosclerosis.

Major surgery induces a surgical stress response that initiates a catabolic metabolism. Furthermore, the risk of systemic inflammatory response syndrome (SIRS) both before and after amputation is high (3) as the most prominent indication for amputation is gangrene, followed by non-healing or infected wounds. This leads to an impaired immune response and an increased insulin resistance that also includes a cascade of impaired appetite regulation, low dietary intake and reduced nutrient uptake form the intestine which increases inflammation, loss of muscle and risk of severe complications.

Among healthy adults with a normal weight a slow speed of eating will result in a low nutritional intake due to faster satiety experience.

Low appetite following major surgery is related to the regulation of hormone controlling the appetite. Especially older patients experience variations in appetite that affect their eating pattern such as eating speed and intake. It is therefore reasonable to assume that the speed of eating and the total nutritional intake among older patients, who are exposed to catabolic metabolism, are associated.

The hypothesis is that major surgery induces a change in patients' current eating pattern that is measurable and can be identified as a surrogate measurement of the catabolic state that is related to inflammation.

Eating Patterns are often described in clinical practice without engaging in nutritional assessment of the patient. Whether the speed of eating is an objective marker of the current nutritional status has not been established.

This study investigates patients undergoing lower limb amputation and their nutritional status, eating pattern and inflammation and whether this is linked to the current degree of disease. The purpose is to describe the development in nutritional status before and after amputation and to investigate associations between patients eating pattern and nutritional status to inflammatory and metabolic biomarkers reflecting the degree of disease.

DETAILED DESCRIPTION:
The study is an observational cohort study that includes patients with lower limb amputation from admission to discharge.

Patients are admitted to a special amputation-unit from the outpatient clinic, the emergency department or other departments at the hospital. All patients with lower limb amputation are treated according to a rehabilitation programme that includes a multidisciplinary approach and a well-defined treatment for pain, fluid, nutrition and mobilisation.

All patients receive a standardised house diet prepared in the hospital kitchen. The diet consists of 18% protein, 40% lipids and 42% carbohydrate. The house diet is supplemented with minimum three in-between meals prepared in the dietary kitchen. The use of protein supplement is also available. Patients´ food and fluid intake are monitored daily.

Data on nutrition and eating pattern

The eating pattern is measured using a digital weight that measure gram per second. The weight is linked to a raspberry computer that recodes all output from the weight. The recording start just before the plate is placed on the weight and ends when the meal is completed. To measure appetite and hunger an arbitrary VAS scale is used to evaluate the patients´ current desire to eat, how hungry they are, how full they fell, and if they want to eat more.

The patients´ nutritional status is evaluated using Mini Nutritional Assessment (MNA). MNA is a valid tool to assess the risk of undernutrition among older people. The MNA consists of a screening tool (max 14 points, < 11 indicates risk of undernutrition) and an evaluation tool (max 16 points). A total point < 23,5 indicates a need for nutritional therapy.

The patients´ behaviour regarding eating and food are evaluated using Eating Identity Type Inventory (EITI). EITI consists of 8 statements that are evaluated by 5 levels of agreement.

The patients´ appetite is evaluated using Simplified nutritional Appetite Questionnaire (SNAQ). SNAQ is a tool validated to evaluate older patients´ appetite. SNAQ consists of four questions with five possible answers with a max score of 20 points. A score <14 points indicates risk of weight loss of 5 %.

Data on Inflammation and metabolism To describe any change in inflammation or metabolic status, serum and plasma samples will be collected after inclusion, on the day of surgery and on 1, 3, 5, and 10 postoperative day. A total of 350 ml blood will be collected over a period of 12 days. The analysis is expecting to consist of inflammatory and metabolic biomarkers. All samples will be contained at minus 80 degree and minus 135 degree for immucells.

The degree of diseases will be measured using the biomarker suPAR that is associated with the degree of disease, LOS and mortality. A clinical difference is 2-3 ng/ml.

Data on protein metabolism To evaluate the protein metabolism, 10 patients undergoing above ankle amputation will have a bladder catheter inserted on the day of surgery, to collect a 24-hour urine sample. The catheter will hereafter be removed. This will be done on the 1, 5, and 10 postoperative day.

Demographic and baseline data Data on patients´ sex, age, marital status, residence, functional mobility, comorbidities, smoking and alcohol use, medications, educational and working status, and use of homecare services will be collected. The patients´ muscle strength is measured using handgrip strength on the dominant hand prior to surgery and on the 5, 10 postoperative day and at discharged.

Complications Complications during hospitalisation will be registered and categorised as; cardio or respiratory, metabolic, infection and lack of healing, re-amputation or revision within 30 days, and 30 day mortality.

The analysis of data will include an investigation of: whether suPAR is dependent on nutritional intake whether; patients' eating pattern can be used as an objective description of the current nutritional status; inflammation is dependent on nutritional intake; complications are dependent on nutritional intake. We will also investigate protein metabolism after lower limb amputation.

Power calculation The aim of the study is to describe the associations between the patients eating pattern and nutritional status and the degree of disease among older patients undergoing lower limb amputation.

We calculated that; with a power of 80%; a statically significant level of 5%; a minimum difference in suPAR at 2,5ng/ml between patients who receive sufficient nourishment or not (assuming that 50% of all patients achieve sufficient nourishment during hospitalisation) and a SD at 2.8 ng/ml (suPAR) the number of included patients should be 42. An estimated dropout set at 20 % (8 patients) results in a inclusion of 50 patients.

The primary outcome is a change in suPAR, a biomarker related to the degree of disease, hospitalization and death. The outcome will be measured before and 10 days after surgery.

The secondary outcomes are; nutritional intake measured as daily protein (g/kg) and energy (kilojoule/kg) intake, eating rate measured as g/min, total length of the meal, activity (activity on the plate compared with intake), biomarkers for inflammation and metabolism; protein balance measured as urine urea nitrogen in a 24-hour urine sample; revisions and re-amputation; LOS and 30 day mortality.

ELIGIBILITY:
Inclusion Criteria:

* Having a medical indication for amputation
* Admitted with a non healing wound on lower limb
* Revision following previous amputation
* Able to speak and understand Danish - able to give an informed consent

Exclusion Criteria:

* Traumatic or pathologic indication for amputation
* Any or current use of narcotics
* Major surgery within the last four weeks
* If not amputated two weeks after admission

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are included from a cohort of patients who are admitted to the Department of Ortopedic Surgery.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2015-08-19 (Actual); Primary Completion 2016-11-13 (Actual); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
suPAR | From admission to ten days after surgery
  Soluble urokinase plasminogen activator receptor: Biomarker of low-grade inflammation. suPAR are measured prior to surgery and on the 1, 3, 5 and 10 postoperative day and will be compared to patients daily intake of energy (kilojoule) and protein (gram)

SECONDARY OUTCOMES:
Inflammatory biomarkers such as IL6, IL10,IL18, TNF-a, MCP-1, sCD14, C reactive protein, expression of inflammatory genes from immucell | From admission to ten days after surgery
  Biomarkers of low-grade inflammation. Inflammatory biomarkers will be measured in duplicates in serum or plasma using commercially available Luminex or ELISA kits according to the manufactures instructions. Cytokines with low systemic levels such as IL-6 and TNF-α will be measured with high sensitive kits to ensure detection. Samples are stored in a biobank established for the project at -80°C. Inflammatory biomarkers are measured simultaneously when all patients have been included.
Metabolic biomarkers such as Insulin, Glucose, Adiponectin, Leptin, Ghrelin | From admission to ten days after surgery
  Biomarkers of metabolic pathway Glucose is measured in blood at each visit using the HemoCue® system. All other metabolic biomarkers will be measured in duplicates in serum or plasma using commercially available Immulite, Luminex or ELISA kits according to the manufactures instructions. Samples are stored in a biobank established for the project at -80°C. Metabolic biomarkers except for glucose are measured simultaneously when all patients have been included.
Postoperative LOS from surgery to medical stability (planned disharge) | From surgery to discharge
  The LOS are measured from the admission day to the unit and to the day the patients medical treatment are completed
Revisions or re-amputation | From surgery to discharge
  A Revision after amputation is defined as a surgical invasive procedure that aims to improve healing of the stump. A re-amputation is also defined as a surgical invasive procedure that includes amputation on a higher level
Severity of Infections | From surgery to discharge
  Infections are categorised in; sepsis, deep wound infections that is treated with antibiotics and superficially wound infections.
Eating patterns (eating time, intake ) | From surgery to ten days after surgery
  Eating pattern are measured as speed of eating (gram per minutes), the time for the total meal (minutes) and total intake (gram).
Secondary analysis 1: Descriptions of the nutritional status during hospitalisation 2: Nutritional status at disharge, dependency of morbitity | 1: From admission to 10 postoperative day 2: Nutritional status at discharge
  1. Nutritional intake is measured in protein (gram) and energy (Kilojoule). The nutritional intake is monitored daily from inclusion to 10 postoperative day.
  2. The nutritional status at discharge measured as difference in bodyweight from admission. Morbidity are defined as any chronical disease registered using ICG 10 code
Protein metabolism | Will be mesured on the 1, 5, and 10 postoperative day
  Analysis of 24 hour urine sample among 10 patients undergoing major lower limb amputation. The protein metabolism will be measured as U-Carbamide (mmol) that are converted to the level of nitrogen and then compared to the daily protein intake to estimate the balance of protein.
Monocytic Myeloid-derived Suppressor Cells (mMDSCs) | Measured at inclusion, and at day 10 after amputation, and at inclusion for Controls
  mMDSC are measured by FACS analyses in cryopreserved peripheral blood mononuclear cells
Sirtuin 1 (SIRT1) | Measured in muscle biopsies taken in the beginning of the amputation for patients, and at inclusion for Controls
  SIRT1 along with other factors regulating hypoxia, inflammation, and catabolism such as hypoxia-inducible factor (HIF)-1a, nuclear factor k B (NF-kB), and forkhead box protein (Fox) O1 are measured in muscle biopsies from patients and controls. Muscle biopsies are submerged in All Protect (Quiagen) immediately after acquisition, and stored at least overnight, before transferral to a new cryo-vial. Muscle biopsies are stored at -80C until analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Ove Andersen, PHD,MD, Principal Investigator — Clinical Research Centre, University Hospital of Copenhagen, Hvidovre
Locations (1):
- University Hospital of Copenhagen, Hvidovre, Hvidovre, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided